CLINICAL TRIAL: NCT06939075
Title: Role of Cross Sectional Imaging Modalities in the Diagnosis and Characterization of Colonic Masses
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maram Kamal Ahmed, ROLE OF Cross sectional imaging modalities in the diagnosis and characterization of colonic masses, Assiut University
Other Study IDs: Diagnosis of colonic masses
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: ROLE OF Cross Sectional Imaging Modalities in the Diagnosis and Characterization of Colonic Masses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: ROLE OF Cross sectional imaging modalities in the diagnosis and characterization of colonic masses — Study tools (in detail, e.g., lab methods, instruments, steps, chemicals, …):
  * CT Scan: To evaluate mass morphology, size, and lymph node involvement.
  * MRI: To assess tissue composition, characterization and diffusion restriction.
  * Colonoscopy and Biopsy: Gold standard reference to assess the diagnostic accuracy for different

SUMMARY:
Colonic masses are frequently encountered in clinical practice and can be benign or malignant. Accurate characterization is crucial for optimal management. Traditional imaging techniques such as colonoscopy remain the gold standard; however, multi-modality imaging-including computed tomography (CT), magnetic resonance imaging (MRI), and positron emission tomography (PET)-has gained importance.

Colorectal cancer (CRC) is one of the most commonly diagnosed malignancies worldwide, ranking as the third most common cancer and the second leading cause of cancer-related mortality. According to the Global Cancer Observatory (GLOBOCAN), in 2020, there were approximately 1.9 million new cases of CRC and over 930,000 deaths. The incidence varies geographically, with higher rates in developed countries due to lifestyle factors, dietary habits, and genetic predispositions. Early detection through screening and imaging plays a pivotal role in reducing morbidity and mortality. (Sung et al., 2021).

Recent studies have demonstrated that multi-modality imaging improves diagnostic confidence in colonic lesions. CT colonography has been shown to have a sensitivity of approximately 96% for detecting polyps ≥10mm (Pickhardt et al., 2019). MRI provides superior soft tissue contrast, aiding in local tumor staging (Beets-Tan et al., 2020). These advancements underline the importance of integrating multiple imaging techniques for comprehensive colonic mass evaluation.

Staging of colorectal cancer is crucial for treatment planning and prognosis assessment. The TNM (Tumor, Node, Metastasis) staging system is widely used:

* T (Tumor size and invasion): Ranges from T1 (tumor confined to the mucosa) to T4 (tumor invading adjacent structures).
* N (Lymph node involvement): N0 (no nodal involvement) to N2 (extensive nodal spread).
* M (Distant metastases): M0 (no metastases) to M1 (presence of metastases). Imaging plays a fundamental role in staging. CT is the primary modality for detecting lymph node involvement and distant metastases (Liu et al., 2020). MRI, particularly with diffusion-weighted imaging, provides superior soft-tissue contrast for local staging, especially in rectal cancer (Maas et al., 2019).

Colonoscopy with histopathological biopsy remains the gold standard for diagnosing colonic masses. It allows direct visualization, biopsy sampling, and polyp removal if necessary.

This study aims to evaluate the diagnostic accuracy and clinical utility of these imaging modalities in detecting and differentiating colonic masses.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years) referred for imaging due to suspected colonic mass. Histopathological confirmation is available.

Exclusion Criteria:

* • Patients with contraindications to contrast imaging as sensitivity to contrast media or renal impairment

  * Patient with contraindication for MRI e.g patients having a devices with Para magnetic effect e.g pacemakers and claustrophobia
  * Patients with prior colorectal cancer diagnosis or surgical intervention

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adults (>18 years) referred for imaging due to suspected colonic mass. Histopathological confirmation is available
Sampling Method: Probability Sample
Enrollment: 111 (Estimated)
Dates: Start 2025-07-24 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
• Accuracy, sensitivity, and specificity of imaging modalities in detecting & diagnosis of colonic masses | two years